CLINICAL TRIAL: NCT03456349
Title: A Phase 1b Randomized, Double-blind, Placebo-controlled, Parallel Group, Multi-center Study to Determine the Safety and Tolerability of HTL0018318 in Subjects With Alzheimer's Disease Receiving Standard-of-care
Brief Title: Multi-centre Study of HTL0018318 in Patients as an add-on to Standard-of-care
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nxera Pharma UK Limited (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HTL0018318-202; 2017-000649-34 (EudraCT Number)
Record Dates: First submitted 2018-02-22; First posted 2018-03-07 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low dose (Experimental): HTL0018318
  Interventions: Drug: HTL0018318
- Medium dose (Experimental): HTL0018318
  Interventions: Drug: HTL0018318
- High dose (Experimental): HTL0018318
  Interventions: Drug: HTL0018318
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HTL0018318 — HTL0018318
  Arms: High dose; Low dose; Medium dose
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Multi-centre study of HTL0018318 in patients with Alzheimer's disease as an add-on to standard-of-care

DETAILED DESCRIPTION:
This is a multi-centre study conducted in four countries. A total of 60 subjects with Alzheimer's disease who are on standard-of-care will be enrolled to receive one of 3 active HTL0018318 or placebo for a period of four weeks

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic evidence of Alzheimer's disease according to the 2011 National Institutes of Aging-Alzheimer's Association (NIA-AA) criteria
2. Participants with Alzheimer's disease on stable standard of care

Exclusion Criteria:

1. Presence of illness apart from Alzheimer's disease that could contribute to cognitive dysfunction
2. A current or history of clinically significant suicidal ideation within the past 6 months
3. Subjects who have been on anti-cholinergic and/or anti muscarinic treatment

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events (TEAEs), Safety and Tolerability | Baseline to Day 28

CONTACTS AND LOCATIONS:
Locations (4):
- Syneos, Prague, Czechia
- Syneos, Warsaw, Poland
- Syneos, Bratislava, Slovakia
- Syneos, Barcelona, Spain